CLINICAL TRIAL: NCT04200547
Title: Prospective, Controlled, Randomized, Multicentered, Open-label Study, Comparing 2 Modalities of Follow-up of Patients With Crohn's Disease, Postoperatively Treated With Adalimumab (Immunomonitoring vs Standard Follow-up)
Brief Title: Interest of the Dosage of Adalimumab Serum Levels in Crohn's Disease Patients for Prevention of Postoperative Recurrence
Acronym: ADAPT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment of participants was no longer sufficient to continue the study.
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RECHMPL19_0071; UF 7772 (Other: UH Montpellier)
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: This is a multicenter, interregional, open-label, prospective comparative PHASE III, randomized with a ratio (1:1), with 2 parallel groups (experimental group called "immunomonitoring" and control group called "standard strategy based on clinical and biological activity").
Who Masked: Outcomes Assessor
Masking Description: An endoscopy will be performed on patients of all groups 6 months after the surgery. Endoscopic results will be measured blindly by one assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunomonitoring-based follow-up (Experimental): Post-operative follow-up of Crohn's disease patients will be done through the measurement of the residual rate of the drug adalimumab in the serum.
  Interventions: Other: Immunomonitoring-based follow-up
- Standard follow-up (Active Comparator): Post-operative follow-up of Crohn's disease patients will be based on clinical and biological parameters. This strategy is the standard strategy for post-operative follow-up of Crohn's disease patients.
  Interventions: Other: Standard follow-up

INTERVENTIONS:
Other: Immunomonitoring-based follow-up — Post-operative follow-up of Crohn's disease patients will be done through the measurement of the residual rate of the drug adalimumab in the serum. Patients will receive adalimumab treatment every other week, starting 1 month after the surgery. 3 months after the surgery, serum levels of adalimumab will be measured:
  * If the level is below 5ug/mL, adalimumab treatment will be increased to every other week until the end of the study.
  * If adalimumab level in the serum is above 5ug/mL, the treatment's frequency will be maintained until the end of the study.
  Arms: Immunomonitoring-based follow-up
Other: Standard follow-up — Post-operative follow-up of Crohn's disease patients will be based on clinical and biological parameters. Patients will receive adalimumab treatment every other week, starting 1 month after the surgery. If clinical relapse (CDAI > 220 together with an increase of 70 points) and biological relapse (CRP > 10mg/mL and fecal calprotectin > 100 ug/g) occur, frequency of adalimumab treatment will be increased to once a week.
  Arms: Standard follow-up

SUMMARY:
Study comparing 2 modalities of Crohn's disease patients postoperative follow-up treated with adalimumab (Humira® or biosimilar) : immunomonitoring of adalimumab serum levels versus standard follow-up, which is based on the clinical and biological activity of the disease.

DETAILED DESCRIPTION:
Patients in the experimental arm will have a post-operative follow-up based on the immunomonitoring of serum levels of adalimumab. After ileocolic resection surgery, patients will have a therapeutic optimization of their adalimumab (Humira® or biosimilar) treatment, based on their serum residual rate of adalimumab.

Patients in the control group will receive a standard post-operative follow-up, which is based on clinical and biological recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patient between the ages of 18 and 75
* Use of an effective method of contraception during treatment with adalimumab for women of childbearing age
* Crohn's disease diagnosed according to the criteria defined by the national and international recommendations for at least 3 months
* IIeocolic resection with ileocolic anastomosis and absence of residual macroscopic lesion, or ileocolic resection with transient ostomy and restoration of continuity
* For anti-TNF-naive patients: negative pre-anti TNF balance
* Indication of postoperative treatment for the prevention of recurrence of Crohn's disease (with at least 1 risk factor for recidivism):

  * active smoking (≥ 1 cigarette / day at the time of surgery)
  * hail resection> 50 cm
  * second intestinal resection
  * presence of anoperineal lesions
  * Penetrating impairment (B3 of the Montreal Classification)
  * Biotherapy treatment for more than 6 months before the surgery
* Written and signed consent by the participant and the investigator
* Affiliated person or beneficiary of the social security system.

Exclusion Criteria:

* Intolerance or allergy to adalimumab (Humira® or biosimilar)
* Patients to whom adalimumab (Humira® or biosimilar) is contraindicated
* Intestinal stoma without restoration of continuity
* Pregnant woman (dosage of positive βHCG) or breastfeeding according to article L1121-5 of the french public health law.
* Contraindication or refusal of ileocolonoscopy at 6 months
* Patient who could not be followed regularly for psychological, social or geographical reasons
* Vulnerable people according to article L1121-6 of the french public health law
* Persons subject to legal protection (guardianship, trusteeship) or unable to express their consent according to Article L1121-8 of the french public health law or under the protection of justice according to article L1122.2 of the CSP
* Concomitant participation of the patient in another research involving the human person.
* Patient not affiliated to the social security system (Article L.1121-11).
* Patient unable to sign the consent form
* Immunized patients (with anti-adalimumab antibodies > 10ng / mL and undetectable adalimumab levels, Elisa drug sensitive technique used) for patients already treated with adalimumab (Humira® or biosimilar) before surgery
* Patients in combination therapy with azathioprine, 6-mercaptopurine or methotrexate Post-operative, or treated by another biotherapy (infliximab, vedolizumab, ustekinumab ...)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a Rutgeerts score ≥ i2 | 6 months
  The primary endpoint will be measured by ileocolonoscopy under general anesthesia after standard preparation by PEG with video recording of the examination, carried out by one of the investigators of the study in each center. An ileocolonoscopy 6 months after intestinal resection remains the reference examination for the endoscopic diagnosis of recurrence according to the endoscopic Rutgeerts score (endoscopic recurrence if Rutgeerts score ≥ i2) and allows the adaptation or the introduction of a treatment to limit clinical recurrence at 18 months.

SECONDARY OUTCOMES:
Percentage of patients with clinical recurrence | 3 and 6 months
  Evaluation of the clinical recurrence after surgery . Evaluation based on the CDAI. (clinical recurrence if CDAI ≥ 220 and ≥70 points increase from baseline CDAI), CRP (> 10mg/L) and fecal calprotectin (> 100μg/ g).
Percentage of patients with biological recurrence | 3 and 6 months
  Biological recurrence will be evaluated based on CRP and fecal calprotectin:
  CRP: 10 mg / L threshold to define a biological recurrence. Fecal Calprotectin: 100 μg / g threshold to define a biological recurrence
Percentage of patients with adverse effects | 3 and 6 months
  The practitioner will assess (through a questionnaire) the presence or absence : of joint pain, allergic reactions, autoimmune reaction, complications at the puncture wound, infections, hospitalization .
Rate of adalimumab in the serum | 1, 3, and 6 months
  Adalimumab levels (in μg/mL) will be measured on a blood sample
Rate of anti-adalimumab antibodies in the serum | 1, 3, and 6 months
  Anti-adalimumab antibodies (ng/mL) will be measured on a blood sample only in cases of undetectable adalimumabemia (Elisa Drug-sensitive technique)

CONTACTS AND LOCATIONS:
Overall Officials: Lucile BOIVINEAU, Principal Investigator — Montpellier University Hospital
Locations (1):
- CHU de Montpellier, Montpellier, France